CLINICAL TRIAL: NCT03765216
Title: Efficacy of Tailored Bowel Preparation Strategy: A Randomized Controlled Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President of Qilu Hospital, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2018SDU-QILU-09
Record Dates: First submitted 2018-12-04; First posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Bowel Preparation; Colonoscopy
MeSH Terms: interventions — Polyethylene Glycols

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to group A or B. Participants of group A are given normal bowel preparation, while participants of group B are given personalized regimens according to a predictive model we have established.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: standard group (Active Comparator): Participants are given standard regimen: 2 L Polyethylene Glycol (PEG) regimen.
  Interventions: Drug: 2L Polyethylene Glycol (PEG)
- Group B: tailored group (Experimental): Participants are given personalized regimens for bowel preparation according to the the predictive model( a model which grades patients as low or high risk according to risk factors such as age, body mass index≧ 30 kg/m2, diabetes, constipation, pelvic surgery and tricyclic antidepressants usage).
  Low risk patients are given standard regimen: 2 L Polyethylene Glycol (PEG) regimen; High risk patients are given standard regimen: 4 L Polyethylene Glycol (PEG) regimen.
  Interventions: Drug: 2L Polyethylene Glycol (PEG); Drug: 4L Polyethylene Glycol (PEG)

INTERVENTIONS:
Drug: 2L Polyethylene Glycol (PEG) — Participants in Group A and Low risk patients in group B are given standard regimen: 2 L Polyethylene Glycol (PEG) regimen
  Other Names: Standard
Drug: 4L Polyethylene Glycol (PEG) — High risk patients in Group B will receive 4 L Polyethylene Glycol (PEG) regimen
  Other Names: High dose
  Arms: Group B: tailored group

SUMMARY:
About 30% of patients were reported to suffer inadequate bowel preparation. So, it is desirable to prescribe personalized regimen according to patient's personal characteristics.

DETAILED DESCRIPTION:
Colonoscopy is currently the main approach for detecting mucosal abnormalities in the whole colon. Inadequate bowel preparation is the predominant threaten to the efficacy of colonoscopy.Unfortunately, about 30% of patients were reported to suffer inadequate bowel preparation. In order to improve adequate bowel preparation rate, it is desirable to prescribe personalized regimen according to patient characteristics. We intend to improve adequate bowel preparation rate by deploying tailored bowel preparation strategy. There are many predictive factors of inadequate bowel preparation such as obesity, constipation, abdominal surgery and so on. By recognizing these risk factors of the patients , we can prescribe the patients with higher dose of bowel cleansing regimen to improve bowel preparation quality.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18 or older
* patients undergoing colonoscopy

Exclusion Criteria:

* patients with a history of colorectal surgery
* patients with severe colonic stricture or obstructing tumor
* patients with dysphagia
* patients with compromised swallowing reflex or mental status
* patients with significant gastroparesis or gastric outlet obstruction
* patients with known or suspected bowel obstruction or perforation
* patients with severe chronic renal failure (creatinine clearance<30 ml/min)
* patients with severe chronic renal failure (creatinine clearance<30 ml/min)
* patients with uncontrolled hypertension (systolic blood pressure>170 mm Hg, diastolic blood pressure>100 mm Hg)
* patients with inflammatory bowel disease or megacolon
* patients with dehydration
* patients with dehydration
* patients with pregnancy or lactation
* patients hemodynamically unstable
* patients unable to give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-03-15 (Estimated)

PRIMARY OUTCOMES:
Adequate bowel preparation rates | 2 months
  Adequate bowel preparation rates between 2 groups according to Boston Bowel Preparation Scale (BBPS)

SECONDARY OUTCOMES:
Polyp detection rate | 2 months
  Polyp detection rates between 2 groups

CONTACTS AND LOCATIONS:
Overall Officials: Li Yanqing, PhD,MD, Principal Investigator — Qilu Hospital of Shandong University
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Ji'nan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data of this trial will be shared when necessary